CLINICAL TRIAL: NCT00239915
Title: An 8-week, Double-Blind, Randomized, Multicenter, Flexible-Dose, Placebo-Controlled Pilot Study of Pagoclone in Patients With Persistent Developmental Stuttering Followed by a 52-week Open-Label Extension.
Brief Title: Safety and Efficacy Study of the Investigational Drug Pagoclone, in the Treatment of Persistent Developmental Stuttering (PDS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pharmacology Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRI#600
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2012-05-09 (Estimated); Status verified 2012-05

CONDITIONS: Persistent Developmental Stuttering
MeSH Terms: interventions — pagoclone

INTERVENTIONS:
Drug: Pagoclone

SUMMARY:
This is a research study of the investigational drug, Pagoclone, in the treatment of persistent developmental stuttering (PDS), which includes frequent repetitions or prolongations of sounds or syllables or words, or frequent hesitations or pauses that disrupt the flow of speech. Pagoclone is an investigational drug, so it is not approved by the United States Food and Drug Administration.

ELIGIBILITY:
Inclusion Criteria:

* PDS defined as DSM-IV-TR criteria
* Symptoms starting before age 8
* Total overall score of 18-36 on the SSI-3
* English speaking, with an 8th grade education
* Able to understand and cooperate with study requirements with assistance
* Not pregnant or breastfeeding
* Able to provide consent

Exclusion Criteria:

* No diagnoses of other CNS/Mental health disorders in the last 6 months
* No use of psychotropic medication or other medication for stuttering within 4 weeks prior to screening
* No use of non-medicinal stuttering treatments for 5 months prior to the study
* No use of illicit drugs or opiates of any kind

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2005-04; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Jon F. Heiser, M.D., Principal Investigator — Pharmacology Research Institute
Locations (1):
- Pharmacology Research Institute, Riverside, California, United States